CLINICAL TRIAL: NCT05950893
Title: The Clinical Feasibility and Validity of Simple Measurement of Inspiratory Muscle Pressure Index (PMIvent) to Access Inspiratory Effort During Pressure Support Ventilation
Brief Title: The Clinical Feasibility and Validity of PMIvent to Access Inspiratory Effort During Pressure Support Ventilation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jian-Xin Zhou (Other)
Responsible Party: Sponsor-Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KT2023-032-02
Record Dates: First submitted 2023-07-01; First posted 2023-07-18 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Mechanical Ventilation
Keywords: pressure support ventilation; inspiratory effort; inspiratory muscle pressure index

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): PMI represents the difference between plateau airway pressure and peak airway pressure (plateau - peak) during an end-inspiratory airway occlusion.
  Interventions: Procedure: pressure support level

INTERVENTIONS:
Procedure: pressure support level — Baseline ventilators were set by the principle of keeping VT/PBW at 6-8ml/kg and RR at 20-30 breaths/min and the decision of the responsible ICU physician. After then the fraction of inspired oxygen (FiO2), positive expiratory end pressure (PEEP), trigger sensitivity, and cycle-off criteria remain unchanged. Downward PS level titration was performed from 20 cmH2O to 2 cmH2O at a 2cm H2O interval. Every PS level was maintained for 20 minutes and then three end-inspiratory holdings (2-3seconds) and three end-expiratory holdings were performed. To avoid additional injury to the lung and diaphragm, the airway peak pressure (Ppeak) was limited to 30cmH2O.Inspiratory effort is measured as pressure generated by inspiratory muscles using esophageal pressure monitoring.

SUMMARY:
It is critical to maintain a relatively normal inspiratory effort during pressure support ventilation (PSV), the support level should be adjusted to match the patient's inspiratory effort. The inspiratory muscle pressure index (PMI) can reflect the elastic work of the respiratory system at the end of inspiration and has a significant correlation with inspiratory effort, and it has the outgoing advantages of being non-invasive and easy to obtain. Previous studies on PMI were based on physiological research and experimental conditions (PMIref), which require special pressure monitoring devices and software to collect and measure airway pressure. If PMI is going to be used in clinical practice, it is necessary to find a simple measurement method of PMI to replace PMIref. Most ventilators have airway pressure monitoring and end-inspiratory holding functions, and PMI can be measured by freezing the ventilator screen (PMIvent). The overall aim of this study was to determine PMIvent's clinical feasibility and validity for accessing inspiratory effort during PSV.

DETAILED DESCRIPTION:
The intensity of effort the respiratory system produces after receiving respiratory center drive is referred to as inspiratory effort. It is critical to maintain a relatively normal inspiratory effort during assist mechanical ventilation. During pressure support ventilation (PSV), the support level should be adjusted to match the patient's inspiratory effort.

The inspiratory muscle pressure index (PMI) is an indicator based on airway pressure (Paw), defined as the difference between plateau pressure (Pplat) and airway peak pressure (Ppeak). PMI can reflect the elastic work of the respiratory system at the end of inspiration and has a significant correlation with end-inspiratory muscle pressure (Pmus,ei) and esophageal pressure time product per breath (PTPes). Current studies have shown that PMI is an accurate indicator of inspiratory effort, and it has the outgoing advantages of being non-invasive and easy to obtain.

Previous studies on PMI were based on physiological research and experimental conditions, which require special pressure monitoring devices and software to collect and measure airway pressure. In this investigation, the standard measurement of PMI (PMIref) was the difference between Pplat at one cardiac cycle (0.5-1.2s) following end-inspiratory occlusion (EIO) and Ppeak at EIO. This measurement method can avoid the interference of cardiac artifacts on Paw to the greatest extent. If PMI is going to be used in clinical practice, it is necessary to find a simple measurement method of PMI to replace PMIref. Most ventilators have airway pressure monitoring and end-inspiratory holding functions, and PMI can be measured by freezing the ventilator screen (PMIvent). When obtaining PMIvent, the operator could only select a relatively stationary Pplat by visual inspection, and the cardiac artifacts could not be avoided.

Several additional issues need to be addressed when PMI is going to be used in clinical practice to monitor inspiratory effort in ventilated patients. Is PMI easy to obtain? Can PMIvent replace PMIref? What is the effect of different ventilators on PMIvent measurement? What is the relationship between PMIvent and inspiratory effort? Can PMIvent detect high/low effort? Therefore, the aims of this study were to explore the clinical acquisition rate of PMI, the agreement between PMIvent and PMIref, and the predicted value of PMIvent for inspiratory effort. The overall aim was to determine PMI's clinical feasibility and validity for accessing inspiratory effort during PSV.

ELIGIBILITY:
Inclusion Criteria:

Adult acute respiratory failure patients undergoing mechanical ventilation were screened daily and enrolled 24 hours after switching to PSV mode

Exclusion Criteria:

1. age younger than 18 years old or older than 85 years
2. known pregnancy and parturient
3. chronic occlusive pulmonary diseases
4. gastric, esophageal injury
5. barotrauma
6. diaphragm dysfunction
7. intracranial hypertension and brain stem injury
8. consciousness level decreased (RASS less than -2 scores)
9. Anticipating withdrawal of life support and/or shift to palliation as the goal of care.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-03-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Agreement of PMIvent and PMIref | 3 hours
  The accuracy of PMIvent compared to PMIref was assessed by a Bland-Altman plot for each ventilator.

SECONDARY OUTCOMES:
Correlation of inspiratory effort and PMIvent | 3 hours
  The inspiratory effort is measured as the pressure generated by inspiratory muscles using esophageal pressure monitoring. This study selected Pmus and PTPes per minute as the reference for inspiratory effort.
The predicted value of PMIvent for low/high effort | 3 hours
  The target range for "high" inspiratory effort was defined as Pmus > 10 cmH2O and PTPes per minute > 200 cmH2O·s·min-1, and the target range for "low" inspiratory effort was defined as Pmus < 5 cmH2O and PTPes per minute < 50 cmH2O·s·min-1.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No